CLINICAL TRIAL: NCT03100383
Title: Influence of Medical Nutrition Therapy and Eating Behavior on Gestational Weight Gain in Women With Diabetes
Brief Title: Influence of Medical Nutrition Therapy and Eating Behavior on Gestational Weight Gain
Status: Completed | Type: Observational
Sponsor: Materno-Perinatal Hospital of the State of Mexico (Other)
Responsible Party: Principal Investigator, Hugo Mendieta Zeron, Chief of the Research Department, Materno-Perinatal Hospital of the State of Mexico
Other Study IDs: 038/13
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Weight Gain; Eating Behavior
Keywords: gestational diabetes; Type2 Diabetes
MeSH Terms: conditions — Weight Gain; Feeding Behavior; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the association of the number of medical nutrition therapy (MNT) consultations and eating behavior (cognitive restraint, uncontrolled eating, and emotional eating) with GWG in women with type 2 diabetes mellitus (T2DM) and gestational diabetes mellitus (GDM).

DETAILED DESCRIPTION:
Women in puerperium with known T2DM or GDM diagnosed at the hospital were invited to participate in the study. Gestational diabetes was diagnosed with a 75-g oral glucose tolerance test. Weight (kg) and height (m) were measured using a mechanical column scale (SECA).

The specific dimensions of eating behavior were measured through the 18-item Three-Factor Eating Questionnaire-18 (TFEQ-18).

The Medical Nutrition Therapy (MNT) was offered every 2-4 weeks. This therapy consists of providing a food plan with the following recommendations: limiting carbohydrate intake to 35-45% of total calories calculated as 30 kcal/kg based on pregestational BMI for an ideal weight .

We evaluated the effect of MNT on GWG using a multiple linear regression model

ELIGIBILITY:
Inclusion Criteria:

* Women in puerperium with known T2DM or GDM diagnosed at the hospital.

Exclusion Criteria:

* Women with a twin or other multiple pregnancy, type 1 diabetes mellitus (T1DM), or intolerance to carbohydrates, and those with additional diseases (hypertensive disorders of pregnancy, hyper- or hypothyroidism, lupus, kidney or liver disease).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women in puerperium with known T2DM or GDM diagnosed at the hospital were invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2014-06-01 (Actual); Study Completion 2014-11-30 (Actual)

PRIMARY OUTCOMES:
Gestational Weight Gain (GWG). | 9 months
  GWG was calculated by subtracting the prepregnancy weight from the weight at the end of third trimester (kg).

SECONDARY OUTCOMES:
Eating behavior | 9 months
  The specific dimensions of eating behavior were measured through the 18-item Three-Factor Eating Questionnaire-18.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Mendieta Zerón, PhD., Principal Investigator — Maternal-Perinatal Hospital "Mónica Pretelini Sáenz"

IPD SHARING:
Plan to Share IPD: No